CLINICAL TRIAL: NCT05806996
Title: Magnesium and Bladder Spasms Following Ambulatory Urologic Procedures
Brief Title: A Study of Magnesium and Bladder Spasms Following Ambulatory Urologic Procedures
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Gregory A Nuttall, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 22-006895
Record Dates: First submitted 2023-03-23; First posted 2023-04-10 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Bladder Spasms
MeSH Terms: interventions — Magnesium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Magnesium Group (Experimental): Subjects having urology surgery per standard of care will receive intravenous magnesium during the surgery.
  Interventions: Drug: Magnesium
- Placebo Group (Placebo Comparator): Subjects having urology surgery per standard of care will receive intravenous placebo during the surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Magnesium — Intravenous infusion, load 50 mg/Kg with infusion of 15 mg/Kg/hour
  Arms: Magnesium Group
Drug: Placebo — Equivalent volume of normal saline
  Arms: Placebo Group

SUMMARY:
This research is being done to find out whether intravenous magnesium is effective in the treatment of bladder spasms after urologic surgery.

ELIGIBILITY:
Inclusion Criteria:

- Be undergoing a bladder invasive procedure with or without planned urinary catheter on Mayo Clinic Gonda 7 Outpatient Procedure Center.

Exclusion Criteria:

* Are unable to grant informed consent or comply with study procedure.
* Allergy or known sensitivity to magnesium or Renacidin.
* Expected or high risk of bladder extravasation.
* Ongoing atrial fibrillation prior to surgery.
* Are undergoing emergency surgery.
* Are pregnant.
* Known hypermagnesemia.
* Patients with neuromuscular weakness (e.g., Myasthenia gravis) due to magnesium's muscle weakening effect.
* Patients with myocardial compromise or cardiac conduction defects because of magnesium's anti-inotropic effects.
* Patients with renal insufficiency, glomerular filtration rate less than 30, since Magnesium is eliminated by the kidneys resulting in exaggerated rise in serum magnesium.
* Patients with concomitant use of a calcium channel blocker since magnesium sulfate could act synergistically to suppress muscular contractility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of bladder spasm | Post-operative, approximately 1 hour
  Number of subjects to experience bladder spasms

SECONDARY OUTCOMES:
Incidence of bladder spasm above moderate grade | Post-operative, approximately 4 hours
  Number of subjects to experience bladder spasms above moderate grade
Treatment for bladder spasms | Post-operative, approximately 4 hours
  Number of subjects requiring treatment for bladder spasms
Patient satisfaction | Post-operative, approximately 4 hours
  Assessed using a seven-point Likert scale where 1=strongly dissatisfied, 2=moderately dissatisfied, 3=slightly dissatisfied, 4=neutral, 5=slightly satisfied, 6=moderately satisfied, 7=extremely satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Nuttall, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No